CLINICAL TRIAL: NCT00261729
Title: Prazosin vs. Paroxetine in Combat Stress Symptoms in OIF/OEF Returnees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Peskind, Elaine - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBA-025-05S; 0026; NCT00240201 (obsolete NCT alias)
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Sleep Disorders; Stress Disorders, Post-Traumatic
Keywords: Paroxetine; Prazosin; Sleep Disorders; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Sleep Wake Disorders; Stress Disorders, Post-Traumatic | interventions — Paroxetine; Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): paroxetine
  Interventions: Drug: Paroxetine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo
- 3 (Experimental): prazosin
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Paroxetine — paroxetine 20 mg
  Other Names: Paxil
  Arms: 1
Drug: Prazosin — Prazosin
  Arms: 3
Drug: placebo — placebo capsules
  Arms: 2

SUMMARY:
Evaluate the efficacy and tolerability of the drug prazosin compared to placebo for combat stress-related nightmares, sleep disturbance and overall function in recently combat-exposed returnees from OIF and OEF. To evaluate the effects of the SSRI paroxetine on behavioral symptoms and overall function in this population.

DETAILED DESCRIPTION:
Trauma-related nightmares and sleep disruption that follow combat exposure are distressing and frequently treatment resistant symptoms that impair quality of life and overall function. These symptoms closely resemble core nighttime symptoms of posttraumatic stress disorder (PTSD), and are increasingly recognized in returnees from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF). Prazosin, a generically available brain active alpha-1 adrenergic receptor antagonist, markedly reduced or eliminated combat trauma-related nightmares and sleep disruption in 23 of 25 combat-exposed returnees from OIF at Madigan Army Medical Center (MAMC). The use of prazosin in OIF returnees was based on clinical efficacy of prazosin for trauma-related nightmares, sleep disturbance, and overall function in Vietnam combat veterans with chronic PTSD. The only drugs FDA approved for PTSD are the selective serotonin reuptake inhibitors (SSRIs) sertraline and paroxetine. However, SSRI effectiveness in combat trauma PTSD, especially for nighttime symptoms, remains questionable.

This is a placebo-controlled clinical trial of prazosin vs. the SSRI paroxetine for combat trauma-related nightmares, sleep disturbance, and overall posttraumatic stress disorder (PTSD) clinical severity in OIF/OEF returnees. Both neurobiologic considerations and our preliminary clinical treatment data provide support for the proposed trial. Preclinical and clinical studies suggest a role for increased central nervous system (CNS) adrenergic outflow and/or responsiveness in PTSD pathophysiology. Possible mechanisms include alpha-1 adrenergic receptor-mediated effects on sleep physiology, corticotropin releasing hormone secretion, and disruption of cognitive processing.

Here we propose a double-blind, placebo-controlled parallel group 12 week clinical trial of prazosin vs. paroxetine to test the following hypotheses:Hypothesis 1. Prazosin will be more effective than paroxetine or placebo for reducing frequency and intensity of combat trauma-related nightmares (as measured by the "distressing dreams" item of the Clinician Administered PTSD Scale [CAPS]).

Hypothesis 2. Prazosin will be more effective than paroxetine or placebo for improving sleep quality (as measured by the Pittsburgh Sleep Quality Index [PSQI]).

Hypothesis 3. Prazosin will be more effective than paroxetine or placebo for improving overall clinical status (as measured by the Clinical Global Impression of Change [CGIC]).

Hypothesis 4. Prazosin will be better tolerated than paroxetine as measured by days retained in the study and frequency of adverse events. Primary outcome measures will assess trauma-related nightmares, sleep disturbance and change in global clinical status: these will include the CAPS [59] Recurrent Distressing Dreams item, the PSQI (60) and the CGIC (58) score. Secondary outcome measures will include total CAPS score, the CAPS subscale scores (Reexperiencing/ Intrusions, Avoidance/Numbing, and Hyperarousal), the Nightmare Frequency Questionnaire (NFQ), Insomnia Severity Index, and measures of depressive signs and symptoms, quality of life, and number of study days completed.

ELIGIBILITY:
Inclusion Criteria:

* Hazardous duty in Iraq or Afghanistan with the US Armed Forces during Operations Iraqi Freedom and Operation Enduring Freedom
* Exposure to at least a moderate level of combat (>5 on Revised Combat Exposure Scale)
* Good general medical health
* Stable dose of non-excluded medications for at least 4 weeks prior to randomization
* >5 on CAPS recurrent distressing dreams item
* >5 on CAPS difficulty falling or staying asleep item

Exclusion Criteria:

* Acute or significant chronic medical illness, preexisting hypotension or orthostatic hypotension, pancreatitis, gout, M ni re's disease, benign positional vertigo, narcolepsy, or any other unstable medical condition.
* Women of childbearing potential with either positive pregnancy test or refusal to use effective birth control method will be excluded.
* Lifetime schizophrenia, schizoaffective disorder, bipolar disorder, psychotic disorder or any DSM-IV cognitive disorder, current delirium, substance dependence disorder within 3 months of the study, severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others.
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist or paroxetine or any other SSRI, no concurrent use of another alpha-1 antagonist agent, no concurrent use an antidepressant (other than trazodone prescribed for sleep).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
CAPS recurrent distressing dreams item | baseline, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | baseline, 6 weeks, 12 weeks
Clinical Global Impression of Change | baseline, 6 weeks, 12 weeks
Total CAPS | baseline, 6 weeks, 12 weeks
Quality of Life Inventory | baseline, 6 weeks, 12 weeks
Penn Alcohol Craving Scale | baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Peskind, MD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Background] Raskind MA, Dobie DJ, Kanter ED, Petrie EC, Thompson CE, Peskind ER. The alpha1-adrenergic antagonist prazosin ameliorates combat trauma nightmares in veterans with posttraumatic stress disorder: a report of 4 cases. J Clin Psychiatry. 2000 Feb;61(2):129-33. doi: 10.4088/jcp.v61n0208. PMID 10732660
- [Background] Peskind ER, Bonner LT, Hoff DJ, Raskind MA. Prazosin reduces trauma-related nightmares in older men with chronic posttraumatic stress disorder. J Geriatr Psychiatry Neurol. 2003 Sep;16(3):165-71. doi: 10.1177/0891988703256050. PMID 12967060
- [Background] Raskind MA, Peskind ER, Kanter ED, Petrie EC, Radant A, Thompson CE, Dobie DJ, Hoff D, Rein RJ, Straits-Troster K, Thomas RG, McFall MM. Reduction of nightmares and other PTSD symptoms in combat veterans by prazosin: a placebo-controlled study. Am J Psychiatry. 2003 Feb;160(2):371-3. doi: 10.1176/appi.ajp.160.2.371. PMID 12562588
- [Background] Raskind MA, Thompson C, Petrie EC, Dobie DJ, Rein RJ, Hoff DJ, McFall ME, Peskind ER. Prazosin reduces nightmares in combat veterans with posttraumatic stress disorder. J Clin Psychiatry. 2002 Jul;63(7):565-8. doi: 10.4088/jcp.v63n0705. PMID 12143911
- [Result] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655
- [Result] Raskind MA, Peskind ER, Hoff DJ, Hart KL, Holmes HA, Warren D, Shofer J, O'Connell J, Taylor F, Gross C, Rohde K, McFall ME. A parallel group placebo controlled study of prazosin for trauma nightmares and sleep disturbance in combat veterans with post-traumatic stress disorder. Biol Psychiatry. 2007 Apr 15;61(8):928-34. doi: 10.1016/j.biopsych.2006.06.032. Epub 2006 Oct 25. PMID 17069768